CLINICAL TRIAL: NCT06859138
Title: Effectiveness of Manual Therapy Added to Splint Therapy Compared to Splint Therapy Alone in the Treatment of Temporomandibular Disorders in Patients Intended for Orthodontic Treatment: a Randomized Clinical Trial
Brief Title: Effects of Occlusal Splint vs Occlusal Splint Added to Manual Therapy in Patients With Temporomandibular Disorders
Acronym: MTvsOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Alfonso Javier Ibáñez-Vera, PhD IN Physiotherapy, Full Professor, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MTvsOS
Record Dates: First submitted 2025-02-23; First posted 2025-03-05 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Temporomandibular Disorders (TMD)
Keywords: temporomandibular disorders; manual therapy; splint therapy; occlusal splint
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Manual therapy and splint therapy (Experimental): Intervention based on manual therapy techniques and splint therapy
  Interventions: Other: Manual Therapy; Other: Splint therapy
- Splint therapy alone (Active Comparator): Intervention based on splint therapy
  Interventions: Other: Splint therapy

INTERVENTIONS:
Other: Manual Therapy — Manual therapy techniques including massage, trigger point pressure, muscle stretching and joint mobilization.
  Arms: Manual therapy and splint therapy
Other: Splint therapy — Dental splint used for temotoromandibular disorders treatment

SUMMARY:
A randomized clinical trial evaluates physiotherapy plus splint treatment versus conventional splint treatment in patients with myofascial-origin temporomandibular disorder (TMD). The study follows the ethical principles of the Declaration of Helsinki and has been approved by the Research Ethics Committee of the University of Jaén.

Methodology Participants, recruited from three dental clinics in Spain, must be adults diagnosed with TMD according to the Diagnostic Criteria for Temporomandibular Disorder (DC/TMD). Patients with health conditions that could hinder participation are excluded. They are randomly assigned to two groups: one receiving physiotherapy plus a splint, and the other receiving only a splint.

The sample size was calculated using G*Power, determining that at least 38 patients (19 per group) are required.

Assessments and Measurements Sociodemographic variables include age, sex, BMI, education level, and lifestyle habits. Various instruments are used to assess TMD and pain, such as the DC/TMD, the Fonseca Anamnestic Index, the Numerical Pain Rating Scale, and the Neck Disability Index.

Intervention Physiotherapy + splint group: Four 20-minute manual therapy sessions, including techniques for the temporomandibular joint and cervical muscles.

Splint-only group: Only splint use as prescribed by the dentist. Assessments are conducted before and after treatment for the physiotherapy group and at two time points for the splint-only group (before splint placement and one month later).

Data Analysis SPSS and MedCalc software will be used, with a 95% confidence level. Relationships will be analyzed through regression and Pearson correlation, and group comparisons will be performed using repeated measures ANOVA, Student's t-test, and Chi-square test. Effect size will be calculated using Cohen's d.

In conclusion, the study aims to determine the effectiveness of combined physiotherapy and splint treatment compared to splint-only treatment in patients with myofascial TMD.

DETAILED DESCRIPTION:
A randomized clinical trial of TM treatment has been designed on patients with TMD of myofascial origin susceptible to dental treatment, complying with the ethical principles for biomedical research in humans formalized in the Declaration of Helsinki. The study has been approved by the Research Ethics Committee of the University of Jaén.

SUBJECTS Subjects are duly informed and their acceptance to participate is formalized by signing an informed consent document where they are also asked for permission to use their photos for the study. Participants are recruited from the Nogales Orthodontic Clinic in Úbeda, the Javier Ruiz Sequera Dental Clinic in Torreperogil, and the SM Medicodental Clinic in Úbeda, Spain. Subjects of legal age affected by myofascial TMD are included, with the diagnosis made using the Diagnostic Criteria for Temporomandibular Disorder (DMD). On the other hand, patients who are not in good physical condition are excluded. The participants were not qualified to understand or carry out the study. The selected participants were randomised into two groups using the Epidat 3.1 software (Conselleria de Sanidade, Xunta de Galicia, Spain), and assigned to a treatment group with physiotherapy plus a splint or another with a conventional approach prescribed with a splint by their dentists.

CALCULATION OF SAMPLE SIZE The sample size was calculated using the G*Power software (latest version 3.1.9.7; Heinrich-Heine University of Düsseldorf, Düsseldorf, Germany) based on the data provided by De Resende et al. A two-tailed hypothesis was considered, 95% power, a p value of 0.05 and an effect size on the VAS of 0.27. A correlation between repeated measures of 0.5 and an effect size of 0.25 were also considered. Taking into account three assessments of the study variables and two study groups, the present study should include a total sample size of at least 38 patients, 19 per group.

MEASUREMENTS All measurements are performed by a trained physiotherapist, who will not know which group each patient belongs to.

The sociodemographic variables taken are age, sex, height, BMI, educational level, whether they work, smoking habits, alcohol habits and physical activity.

Tests and questionnaires:

As for TMD, it is assessed using the DC/TMD, the 'gold standard' test for the diagnosis of TMD, although it is also assessed with the Fonseca Anamnestic Index: a questionnaire made up of 10 questions that can be answered as yes, no and sometimes with a score range between 0 and 100 points.

In addition, pain perception is assessed using the Numerical Pain Rating Scale, a test that grades pain between 0 and 10. In this study, the researchers used this test to assess TMD and neck pain.

To assess neck function, the researchers used the Neck Disability Index, a 10-item questionnaire that provides information on how neck pain has affected the ability to manage daily life.

INTERVENTION The treatment protocol for the physiotherapy plus splint group consists of 4 sessions of 20 minutes each of manual therapy that includes the manual techniques found in the previous systematic review: TMJ articulation, intraoral therapy for the pteregoid muscles, manual therapy for the masseter and temporal muscles, treatment of trigger points with ischemic pressure, and manual therapy for the muscles of the cervical region, sternocleidomastoid, suboccipital, and trapezius.

The treatment protocol for the control group consists of only the use of the splint as prescribed by the dentist. The assessments of the subjects in the physiotherapy plus splint group are carried out before and after each treatment, which will be repeated one week, one week after the latter, and one week after this. The assessments of the subjects in the control group will be carried out before placing the splint and one month after it.

DATA ANALYSIS Statistical analysis will be performed with a confidence level of 95% (p<0.05) and the statistical packages SPSS 19.0 and MedCalc 14.12.043 will be used. Continuous variables will be described by means and standard deviations and categorical variables with frequencies and percentages. The Kolmogorov-Smirnov test will be used to observe the normality of the distribution of the groups. The relationships between the variables will be analyzed by regression and Pearson correlation. Cohen's d will be calculated to measure the effect size in the bivariate analysis and will be calculated as the difference in measurements between the groups divided by the pooled standard deviation of both groups. Cohen's d can be interpreted as the effect size; if the result is 0.2 or less the effect is insignificant, between 0.2 and 0.5 the effect size is small, between 0.5 and 0.8 the effect is medium and a value greater than 0.8 the effect is large. For comparison of the two groups of patients, the Student t-test and the Chi-square test will be used.

Comparisons between the physiotherapy plus splint treatment group and the splint treatment group will be made using a repeated measures analysis of variance (ANOVA), followed by Bonferroni to compare the replicate means for the time points investigated.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with myofascial temporomandibular disorders according to DC/TMD criteria.
* Participants over 18 years old (local legal age).

Exclusion Criteria:

* Participants unable to understand the questionnaires and assessments required for the study due to any condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2025-03-06 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Self reported Temporomandibular Functionning | From the enrollment to end of treatment at one month
  -Fonseca Anamnestic Index: self reported questionnaire about tamporomandibular symptoms.
Mouth opening | From enrollment to the end of treatment at one month
  Maximum mouth opening in millimeters
Temporomandibular functioning | From enrollment to the end of treatment at one month
  -Helkimo Clinical Dysfunction Index: temporomandibular symptoms index to be fulfilled by evaluator.

SECONDARY OUTCOMES:
Cervical function | From enrollment to the end of treatment at one month
  Neck Disability Index, questionnaire measuring cervical functioning or disability
Pain in temporomandibular joint | From enrollment to the end of treatment at one month
  Temporomandibular pain felt by the participant measured with numerical pain rating scale (scores from 0 (no pain) to 10 (higher pain))
Headache or Cephalea | From enrollment to the end of treatment at one month
  Self-reported headache symptoms measured with Head Impact Test questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Villa Aragón, Úbeda, Spain, Spain

IPD SHARING:
Plan to Share IPD: Yes
The data of the study will be available under reasonable request to the corresponding author or published in the Repository of the university of Jaen (www.ruja.es)
Supporting Information: Study Protocol, SAP, CSR
Time Frame: From the publication of the manuscript about the study report until with no end date.
Access Criteria: Any request by email will be attended, as well as everybody could access to RUJA repository as it is public. For access, people will have to request by email or access to www.ruja.es
URL: https://ruja.ujaen.es/home

REFERENCES:
- [Background] Villar-Aragon-Berzosa V, Obrero-Gaitan E, Lerida-Ortega MA, Lopez-Ruiz MDC, Rodriguez-Almagro D, Achalandabaso-Ochoa A, Molina-Ortega FJ, Ibanez-Vera AJ. Manual Therapy Techniques Versus Occlusal Splint Therapy for Temporomandibular Disorders: A Systematic Review with Meta-Analysis. Dent J (Basel). 2024 Nov 1;12(11):355. doi: 10.3390/dj12110355. PMID 39590405
- [Background] Oliveira-Campelo NM, Rubens-Rebelatto J, Marti N-Vallejo FJ, Alburquerque-Sendi N F, Fernandez-de-Las-Penas C. The immediate effects of atlanto-occipital joint manipulation and suboccipital muscle inhibition technique on active mouth opening and pressure pain sensitivity over latent myofascial trigger points in the masticatory muscles. J Orthop Sports Phys Ther. 2010 May;40(5):310-7. doi: 10.2519/jospt.2010.3257. PMID 20436241
- [Background] La Touche R, Fernandez-de-las-Penas C, Fernandez-Carnero J, Escalante K, Angulo-Diaz-Parreno S, Paris-Alemany A, Cleland JA. The effects of manual therapy and exercise directed at the cervical spine on pain and pressure pain sensitivity in patients with myofascial temporomandibular disorders. J Oral Rehabil. 2009 Sep;36(9):644-52. doi: 10.1111/j.1365-2842.2009.01980.x. Epub 2009 Jul 14. PMID 19627454